CLINICAL TRIAL: NCT07253857
Title: Effects of Hand and Arm Bimanual Intensive Therapy Including Lower Extremity on Motor Function and Cognition in Children With Spastic Cerebral Palsy
Brief Title: Effects of Hand and Arm Bimanual Intensive Therapy Including Lower Extremity in Spastic Cerebral Palsy
Acronym: HABIT-ILE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/039 Aleena
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy; Cerebral Palsy, Spastic
Keywords: HABIT-ILE; Intensive motor therapy; Cerebral Palsy; diplegic cerebral palsy with spasticity; Spastic cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: After recruitment into study the participants will be allocated into their respective groups utilizing the online randomizer tool.
Who Masked: Outcomes Assessor
Masking Description: Single blinding approach will be utilized only outcome accessor will be blinded of the allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP -A HABIT-ILE Therapy (Experimental): Name of intervention : Hand and Arm Bimanual Intensive Therapy Including Lower Extermity Type of intensity; intensive , activity based camp style rehabilitation program The HABIT-ILE therapy sessions will be structured to target both upper and lower limbs divided into three categories. Half of each session will focus on table-based bimanual tasks with postural challenges, performed while sitting on fitness balls or standing on balance boards to progressively increase trunk and balance control. Children will practice activities such as drawing, puzzles, crafts, and object manipulation using both hands. About one-third of the session will involve activities of daily living in standing or walking positions, including dressing, grooming, carrying trays, and retrieving items, encouraging functional mobility and postural adaptation. The remaining portion will emphasize gross motor play, such as bowling and ball games, to promote symmetrical movement and coordination.
  Interventions: Other: GROUP -A , Hand and Arm Bimanual Intensive Therapy Including Lower Extremity
- GROUP- B Conventional Physical Therapy (Experimental): The intervention will be delivered five times per week, with each movement repeated three to five times. Sessions will begin at low to moderate intensity and will gradually progress based on patient response. Exercises will include weight-bearing activities such as sit-to-stand transitions to strengthen quadriceps and gluteal muscles, step initiation drills to activate tibialis anterior and gastrocnemius for proper foot placement, and reaching tasks with trunk activation to improve core and upper limb strength. Additional activities will involve lateral and facilitated weight shifts to enhance hip abductor function and postural stability, trunk activation for balance, slow rhythmic movements to manage tone, and controlled handling to reduce spasticity.
  Cognitive therapy will be provided four times per week, lasting about 15 minutes per session. Tasks will initially focus on engagement and stimulation, progressing in complexity.
  Interventions: Other: GROUP-B , Conventional Physical Therapy

INTERVENTIONS:
Other: GROUP -A , Hand and Arm Bimanual Intensive Therapy Including Lower Extremity — Hand Arm Bimanual Intensive Therapy Including Lower Extremity being a task based intensive therapy activities will be structured according to the participants ability to preform it. The intervention incorporates structured bimanual activities that progressively increase in motor complexity, along with functional tasks that necessitate coordinated use of both hands, systematically integrating postural and lower-extremity demands.
  Before therapy begins, each child will participate in a baseline assessment, skilled, repetitive UE movements will be encouraged through both whole task practices where child performs the entire movement without breaking it into smaller component (15-30 min) and part task practice (for 30 sec) .The tasks will be modified to include challenges related to lower extremity and bimanual coordination in upper limb.
  Other Names: HABIT-ILE; HABIT-ILE Therapy; Hand-Arm Bimanual Intensive Therapy Including Lower Extremities
  Arms: GROUP -A HABIT-ILE Therapy
Other: GROUP-B , Conventional Physical Therapy — Conventional therapy will include stretches of lower extremity following bobath approach and cognitive exercises.
  Arms: GROUP- B Conventional Physical Therapy

SUMMARY:
Cerebral palsy (CP), particularly the spastic diplegic subtype, is characterized by motor impairments such as spasticity and mobility limitations. In addition to motor dysfunction, children with CP often experience cognitive impairments affecting decision-making, problem-solving, working memory, selective attention, and inhibitory control. These non-motor challenges contribute to reduced social interaction and quality of life.

Hand-Arm Bimanual Intensive Therapy Including Lower Extremity (HABIT-ILE) has demonstrated improvements in gross motor function among children with spastic CP. However, evidence regarding its impact on cognitive outcomes remains limited. This randomized controlled trial (RCT) aims to evaluate the effects of HABIT-ILE compared with conventional therapy on both motor and cognitive functions in children with spastic diplegic CP. By addressing both upper and lower limb the research seeks to provide a comprehensive therapeutic approach that may yield more significant developmental benefits. Ultimately, the findings could inform the interventions for improving outcomes in pediatric populations affected by diplegic cerebral palsy.

Participants will receive 90 hours of intervention, with assessments conducted at baseline, mid-intervention, and post-intervention. The study will investigate outcomes across motor domains and cognitive functions such as inhibitory control and working memory. Findings are expected to inform comprehensive therapeutic approaches to improve developmental outcomes and quality of life in pediatric populations affected by spastic diplegic CP.

DETAILED DESCRIPTION:
Cerebral palsy is a group of permanent movement and posture disorder caused by damage to the developing brain typically before, during or after birth. It is one of the most common neurodevelopmental disorder in childhood. Spasticity accounts for the majority of cases (around 92%), followed by dyskinesia, hypotonia, ataxia, and mixed types. Within spastic CP, three subtypes are recognized: diplegia, quadriplegia, and hemiplegia. Spastic diplegia is defined by bilateral spasticity with greater involvement of the lower limbs than the upper limbs. It leads to the development of motor and non-motor impairments. The underlying pathology typically involves corticospinal tract damage occurring before, during, or shortly after birth, often linked to prematurity, hypoxic events, or neonatal infections. The motor functions limits functional independence in more extent that cognitive functions. The primary focus of cerebral palsy treatment has been on its motor impairments, particularly spasticity and mobility challenges. According to the recent evidence the individuals with spastic diplegia often experience cognitive impairments especially deficits in executive function. There is growing awareness about these cognitive impairments but interventions for managing executive dysfunction in cerebral palsy patients are still lacking.

The rehabilitation strategies for CP traditionally emphasize physical therapy approaches such as Bobath therapy, Rood's method and Task-oriented training. The task-oriented interventions focus on practicing real-life activities to improve functional independence. More recent evidence supports that activity based approaches such as constraint induced movement therapy and goal directed training, which have shown greater effectiveness than traditional neurodevelopmental therapy. These interventions often targets the specific areas such as upper limb function while neglecting broader impairments involving lower extremities and trunk coordination.

The intensive therapy, Hand-Arm Bimanual Intensive Therapy Including Lower Extremity (HABIT-ILE) was developed to address this limitation. HABIT-ILE integrates upper and lower limb training with trunk control in a structured rehabilitation program. It emphasizes playful, repetitive, and progressively shaped voluntary movements to enhance gross motor skills, postural control, and functional independence.

HABIT-ILE is a camp based intervention in which structured tasks are provided to the participants and the intensity of each task is progressed with time. The maximum of 8-12 participants is in included in one camp. Participants will be divided in 2 groups control group (n= 21) and intervention group (n=21) sample size consisting of 42 participants. The intervention will be provided for total of 90 hour for each group. As these children have limited attention span the typical 9 hour/day intervention is reduced to 3 hour/day for 6 weeks, 5 days a week for the intervention group. For the control group the intervention session will last for 1 hour in morning and 1 hour in evening home exercise plan per day for 9 weeks, 5 days a week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diplegic cerebral palsy
* CP children with manual ability level 1-3 on manual ability classification system
* Participants with gross motor function classification system level ranging from 1-3 will be included in the study.
* With an ability to grasp light objects and lift the more affected arm 15 cm above a table surface.
* Base line cognition level should be 20 or above assessed through mini mental state exam for children (MMC).

Exclusion Criteria:

* Uncontrolled seizures
* Recent or planned botulinum toxin injections within 6 months
* Any recent orthopedic interventions that may affect motor function
* Visual impairments impeding with treatment protocol

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure 88 (GMFM-88) | Outcome will be assessed at 3 points Experimental group(HABIT-ILE);assessment will be done at baseline , after 3rd week and than after 6th week. Experimental group(conventional therapy); Outcome will be assesed at base line, after 4.5 weeks and after 9
  It is a standardized assessment tool designed to evaluate motor function in children with cerebral palsy (CP). It consists of 88 items that measure gross motor abilities across five domains: lying & rolling, sitting, crawling & kneeling, standing, and walking, running & jumping. Each domain is scored on a 4-point ordinal scale where 0 indicates the child does not initiate the movement, 1 reflects initiation with less than 10% completion, 2 represents partial completion between 10% and less than 100%, and 3 denotes full completion of the movement as intended. Higher scores means that the child can move more independently while lower scores show difficulties in movement and point to areas where therapy is needed.
Behavior Rating Inventory Of Executive Function-2 (BRIEF-2) Parent form | Outcome will be assessed at 3 points Experimental group(HABIT-ILE);assessment will be done at baseline , after 3rd week and than after 6th week. Experimental group(conventional therapy); Outcome will be assesed at base line, after 4.5 weeks and after 9
  It assesses executive function in children, including those with cerebral palsy (CP), measuring impulse control, emotional regulation, and working memory
ABILOCO-KIDS-CP | Outcome will be assessed at 3 points Experimental group(HABIT-ILE);assessment will be done at baseline , after 3rd week and than after 6th week. Experimental group(conventional therapy); Outcome will be assesed at base line, after 4.5 weeks and after 9
  This assessment tool designed to evaluate locomotion ability in children with cerebral palsy
ABILHAND-KIDS-CP | Outcome will be assessed at 3 points Experimental group(HABIT-ILE);assessment will be done at baseline , after 3rd week and than after 6th week. Experimental group(conventional therapy); Outcome will be assesed at base line, after 4.5 weeks and after 9
  it is an assessment tool designed to evaluate manual ability in children with cerebral palsy. It focuses on bimanual activities, measuring the child's ability to perform daily tasks requiring upper limb coordination.
Box and Block Test (BBT) | Outcome will be assessed at 3 points Experimental group(HABIT-ILE);assessment will be done at baseline , after 3rd week and than after 6th week. Experimental group(conventional therapy); Outcome will be assesed at base line, after 4.5 weeks and after 9
  It is assessment tool for evaluating manual dexterity in individuals with cerebral palsy. It measures gross motor coordination of the upper limbs by assessing the ability to grasp, transport, and release small blocks within a timed period.
6 Minute Walk Test | Outcome will be assessed at 3 points Experimental group(HABIT-ILE);assessment will be done at baseline , after 3rd week and than after 6th week. Experimental group(conventional therapy); Outcome will be assesed at base line, after 4.5 weeks and after 9
  It evaluates how far a person can walk in six minutes

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Principal Investigator — Lahore University of Biological and Applied Sciences
Locations (1):
- Pakistan Society for Rehabilitation of Differently Abled (PSRD), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park EY. Stability of the gross motor function classification system in children with cerebral palsy for two years. BMC Neurol. 2020 May 6;20(1):172. doi: 10.1186/s12883-020-01721-4. PMID 32375677
- [Background] Craig F, Savino R, Trabacca A. A systematic review of comorbidity between cerebral palsy, autism spectrum disorders and Attention Deficit Hyperactivity Disorder. Eur J Paediatr Neurol. 2019 Jan;23(1):31-42. doi: 10.1016/j.ejpn.2018.10.005. Epub 2018 Nov 2. PMID 30446273